CLINICAL TRIAL: NCT04506255
Title: Silicone Taping for the Improvement of Abdominal Donor Site Scars Following Autologous Breast Reconstruction; A Randomized, Prospective Controlled Trial
Brief Title: Silicone Taping for the Improvement of Abdominal Donor Site Scars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Jason Williams, Principal Investigation, Nova Scotia Health Authority
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 1025794
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Hypertrophic Scar; Scar
Keywords: Silicone; Scar; Abdominoplasty; Breast Reconstruction
MeSH Terms: conditions — Cicatrix, Hypertrophic; Cicatrix

STUDY DESIGN:
Intervention Model Description: This is a prospective, single center, masked, randomized self-controlled clinical human trial to evaluate the appearance of abdominal scars after autologous free-flap breast reconstruction following post-operative application of silicone tape to improve scar quality.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Staff surgeons who are responsible for assessing outcomes will be masked to which side is receiving the silicone tape. At the initial two-week post-op visit, patients will meet with the research coordinator for randomization assignments of their incisions. Surgeons will be masked to assignments. Patients will remove their dressings one day prior to their appointment with their surgeon. This will ensure no local reaction (i.e. redness after tape removal) that would compromise the masking of staff surgeons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silicone tape (Experimental): Adult subjects will act as their own control and will be randomized to have silicone tape applied to one half of their abdominoplasty incision. Patients will apply silicone tape on a daily basis, with each piece lasting 24 hours. Tape may be removed for showers and replied after drying. Total length of treatment will be two and a half months.
  Interventions: Device: Silicone tape
- No dressing (No Intervention): Control treatment using the current standard of care at our institution to the other half, which is no dressing after the initial two week post-op period, will be used on the other half of the incision for comparison. Each individual patient will act as their own control.

INTERVENTIONS:
Device: Silicone tape — Medical grade tape with silicone adhesive
  Arms: Silicone tape

SUMMARY:
This study will look at silicone tape compared to the current no dressing standard at the investigators institution, to determine if silicone tape provides a significant improvement in post-abdominoplasty scar appearance. Silicone tape will be added to half of the abdominoplasty incision of patients undergoing abdominally-based breast reconstruction procedures two weeks after their operation. They will be followed up and assessed at specific timepoints to determine whether the silicone improves scar outcomes in these patients.

DETAILED DESCRIPTION:
This is a prospective, single center, masked, randomized self-controlled clinical human trial to evaluate the appearance of abdominal scars after autologous free-flap breast reconstruction following post-operative application of silicone tape to improve scar quality. Incisions from 32 adult subjects will act as their own control and will be randomized to have silicone tape applied to one half of their abdominoplasty incision and control treatment using the current standard of care at the investigators institution to the other half, which is no dressing after the initial two week post-op period. A participant size of 32 leaves room in case of participant loss to follow-up, ensuring data will be available for the required sample size of 28 (see statistical analysis section below). A random number sequence generator will be used to randomize which half of the patient's wound will receive the treatment.

Patients will be recruited from plastic surgery clinics at the Queen Elizabeth II (QEII) Health Sciences Centre in Halifax, Nova Scotia. Plastic surgeons will be asked to participate and enroll their breast reconstruction patients, who will undergo a type of abdominoplasty as part of their reconstruction procedure.

Patients will undergo a de novo abdominoplasty procedure as part of a reconstructive breast surgery. Two weeks post-operatively, one side of the patient's abdominoplasty incision will be randomized to receive the silicone tape and the remaining half will be left to heal without any dressing application, which is the current standard at the investigators institution. Each patient will act as their own control. Patients will apply silicone tape on a daily basis, with each piece lasting 24 hours. Tape may be removed for showers and replied after drying. Total length of treatment will be two and a half months.

It is not possible to mask patients, as they will be responsible for ongoing application of the silicone tape. However, the staff surgeon will be masked. Patients will present to their first post-op visit at two weeks. After examination by the staff surgeon, the patient will be seen by the research coordinator who will provide the patient with their randomization treatment assignment. To ensure ongoing masking, at subsequent follow-up visits, patients will remove their dressings one day prior to their appointment with their surgeon. This will ensure no local reaction (i.e. redness after tape removal) that would compromise the masking of staff surgeons.

Patients will then follow up for scar assessment at 6 weeks, 3 months, 6 months and 12 months. Unless otherwise required, scar assessments will then be performed at each visit by both the patient and the surgeon using validated objective and subjective scar measures. Patients will also meet with the research coordinator at each follow up visit, to address any questions or concerns about the study and treatment.

The Patient and Observer Scar Assessment Scale (PSAS & OSAS) system will be used to measure scar appearance. The PSAS and OSAS are tools that the patient uses to assess the scar on color, irregularity, itch, pain, thickness, stiffness and overall opinion, and the surgeon uses to assess pigmentation, pliability, relief, surface area, thickness, vascularity and overall opinion (Appendix A). Of note, only the sum of the components of the OSAS portion of the assessment scale is included to calculate the power and sample size, and will therefore be the primary outcome. Secondary outcomes will include the sum of the components of the PSAS score and the overall scores out of 10 for both the PSAS and OSAS from the patient and masked surgeon.

ELIGIBILITY:
Inclusion Criteria:

* undergoing de novo abdominoplasty procedures as part of their breast reconstruction

Exclusion Criteria:

* patients with a history of collagen disease, connective tissue disorders, psoriasis or lupus
* patients with scleroderma
* patients with a history of adverse reaction to adhesives or silicone allergy
* patients with signs of dehiscence or infection resulting in modification to the experimental or control dressings
* patients who are unable to care for their incisions
* patients who are current smokers
* patients who are currently on steroids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale (PSAS & OSAS) System | 6 week follow up, 3 months, 6 months and 12 months.
  The POSAS is a tool that the patient uses to assess the scar on color, irregularity, itch, pain, thickness, stiffness and overall opinion, and the surgeon uses to assess pigmentation, pliability, relief, surface area, thickness, vascularity and overall opinion. Each component is scored out of 10, with a lower score indicating a better scar. Of note, only the sum of the components of the OSAS portion of the assessment scale is included to calculate the power and sample size, and will therefore be the primary outcome.
Patient and Observer Scar Assessment Scale (PSAS & OSAS) System | 3 month follow up
  The POSAS is a tool that the patient uses to assess the scar on color, irregularity, itch, pain, thickness, stiffness and overall opinion, and the surgeon uses to assess pigmentation, pliability, relief, surface area, thickness, vascularity and overall opinion. Each component is scored out of 10, with a lower score indicating a better scar. Of note, only the sum of the components of the OSAS portion of the assessment scale is included to calculate the power and sample size, and will therefore be the primary outcome.
Patient and Observer Scar Assessment Scale (PSAS & OSAS) System | 6 month follow up
  The POSAS is a tool that the patient uses to assess the scar on color, irregularity, itch, pain, thickness, stiffness and overall opinion, and the surgeon uses to assess pigmentation, pliability, relief, surface area, thickness, vascularity and overall opinion. Each component is scored out of 10, with a lower score indicating a better scar. Of note, only the sum of the components of the OSAS portion of the assessment scale is included to calculate the power and sample size, and will therefore be the primary outcome.
Patient and Observer Scar Assessment Scale (PSAS & OSAS) System | 12 month follow up
  The POSAS is a tool that the patient uses to assess the scar on color, irregularity, itch, pain, thickness, stiffness and overall opinion, and the surgeon uses to assess pigmentation, pliability, relief, surface area, thickness, vascularity and overall opinion. Each component is scored out of 10, with a lower score indicating a better scar. Of note, only the sum of the components of the OSAS portion of the assessment scale is included to calculate the power and sample size, and will therefore be the primary outcome.

SECONDARY OUTCOMES:
Patient and Observer Scar Assessment Scale (PSAS & OSAS) System | 6 week follow up
  Secondary outcomes will include the sum of the components of the PSAS score and the overall scores out of 10 for both the PSAS and OSAS from the patient and masked surgeon. A lower score in each component indicates an improved scar.
Patient and Observer Scar Assessment Scale (PSAS & OSAS) System | 3 month follow up
  Secondary outcomes will include the sum of the components of the PSAS score and the overall scores out of 10 for both the PSAS and OSAS from the patient and masked surgeon. A lower score in each component indicates an improved scar.
Patient and Observer Scar Assessment Scale (PSAS & OSAS) System | 6 month follow up
  Secondary outcomes will include the sum of the components of the PSAS score and the overall scores out of 10 for both the PSAS and OSAS from the patient and masked surgeon. A lower score in each component indicates an improved scar.
Patient and Observer Scar Assessment Scale (PSAS & OSAS) System | 12 month follow up
  Secondary outcomes will include the sum of the components of the PSAS score and the overall scores out of 10 for both the PSAS and OSAS from the patient and masked surgeon. A lower score in each component indicates an improved scar.

CONTACTS AND LOCATIONS:
Overall Officials: Jason G Williams, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Halifax Infirmary, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Longaker MT, Rohrich RJ, Greenberg L, Furnas H, Wald R, Bansal V, Seify H, Tran A, Weston J, Korman JM, Chan R, Kaufman D, Dev VR, Mele JA, Januszyk M, Cowley C, McLaughlin P, Beasley B, Gurtner GC. A randomized controlled trial of the embrace advanced scar therapy device to reduce incisional scar formation. Plast Reconstr Surg. 2014 Sep;134(3):536-546. doi: 10.1097/PRS.0000000000000417. PMID 24804638
- [Background] Bleasdale B, Finnegan S, Murray K, Kelly S, Percival SL. The Use of Silicone Adhesives for Scar Reduction. Adv Wound Care (New Rochelle). 2015 Jul 1;4(7):422-430. doi: 10.1089/wound.2015.0625. PMID 26155385
- [Background] Hsu KC, Luan CW, Tsai YW. Review of Silicone Gel Sheeting and Silicone Gel for the Prevention of Hypertrophic Scars and Keloids. Wounds. 2017 May;29(5):154-158. PMID 28570253
- [Background] Sidgwick GP, McGeorge D, Bayat A. A comprehensive evidence-based review on the role of topicals and dressings in the management of skin scarring. Arch Dermatol Res. 2015 Aug;307(6):461-77. doi: 10.1007/s00403-015-1572-0. Epub 2015 Jun 5. PMID 26044054
- [Background] Meaume S, Le Pillouer-Prost A, Richert B, Roseeuw D, Vadoud J. Management of scars: updated practical guidelines and use of silicones. Eur J Dermatol. 2014 Jul-Aug;24(4):435-43. doi: 10.1684/ejd.2014.2356. PMID 25141160
- [Background] Finnerty CC, Jeschke MG, Branski LK, Barret JP, Dziewulski P, Herndon DN. Hypertrophic scarring: the greatest unmet challenge after burn injury. Lancet. 2016 Oct 1;388(10052):1427-1436. doi: 10.1016/S0140-6736(16)31406-4. PMID 27707499
- [Background] Lorenz HP, Adzick NS. Scarless skin wound repair in the fetus. West J Med. 1993 Sep;159(3):350-5. PMID 8236977
- [Background] Gurtner GC, Werner S, Barrandon Y, Longaker MT. Wound repair and regeneration. Nature. 2008 May 15;453(7193):314-21. doi: 10.1038/nature07039. PMID 18480812
- [Background] Mustoe TA. Evolution of silicone therapy and mechanism of action in scar management. Aesthetic Plast Surg. 2008 Jan;32(1):82-92. doi: 10.1007/s00266-007-9030-9. Epub 2007 Oct 30. PMID 17968615
- [Background] Mustoe TA, Cooter RD, Gold MH, Hobbs FD, Ramelet AA, Shakespeare PG, Stella M, Teot L, Wood FM, Ziegler UE; International Advisory Panel on Scar Management. International clinical recommendations on scar management. Plast Reconstr Surg. 2002 Aug;110(2):560-71. doi: 10.1097/00006534-200208000-00031. PMID 12142678
- [Background] O'Brien L, Jones DJ. Silicone gel sheeting for preventing and treating hypertrophic and keloid scars. Cochrane Database Syst Rev. 2013 Sep 12;2013(9):CD003826. doi: 10.1002/14651858.CD003826.pub3. PMID 24030657
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Truong PT, Lee JC, Soer B, Gaul CA, Olivotto IA. Reliability and validity testing of the Patient and Observer Scar Assessment Scale in evaluating linear scars after breast cancer surgery. Plast Reconstr Surg. 2007 Feb;119(2):487-94. doi: 10.1097/01.prs.0000252949.77525.bc. PMID 17230080
- [Background] Fearmonti R, Bond J, Erdmann D, Levinson H. A review of scar scales and scar measuring devices. Eplasty. 2010 Jun 21;10:e43. PMID 20596233
- [Background] Khoo TL, Halim AS, Zakaria Z, Mat Saad AZ, Wu LY, Lau HY. A prospective, randomised, double-blinded trial to study the efficacy of topical tocotrienol in the prevention of hypertrophic scars. J Plast Reconstr Aesthet Surg. 2011 Jun;64(6):e137-45. doi: 10.1016/j.bjps.2010.08.029. Epub 2010 Sep 24. PMID 20869928
- [Background] Kappel S, Kleinerman R, King TH, Sivamani R, Taylor S, Nguyen U, Eisen DB. Does wound eversion improve cosmetic outcome?: Results of a randomized, split-scar, comparative trial. J Am Acad Dermatol. 2015 Apr;72(4):668-73. doi: 10.1016/j.jaad.2014.11.032. Epub 2015 Jan 23. PMID 25619206
- [Background] Joo JS, Zhuang AR, Tchanque-Fossuo C, Tartar D, Armstrong AW, King TH, Sivamani RK, Eisen DB. Dermal suture only versus layered closure: A randomized, split wound comparative effectiveness trial. J Am Acad Dermatol. 2019 Dec;81(6):1346-1352. doi: 10.1016/j.jaad.2019.08.040. Epub 2019 Aug 21. PMID 31442535
- [Background] Duncan JAL, Bond JS, Mason T, Ludlow A, Cridland P, O'Kane S, Ferguson MWJ. Visual analogue scale scoring and ranking: a suitable and sensitive method for assessing scar quality? Plast Reconstr Surg. 2006 Sep 15;118(4):909-918. doi: 10.1097/01.prs.0000232378.88776.b0. PMID 16980850